CLINICAL TRIAL: NCT06278220
Title: Scheimpflug Versus Placido-disc System in Evaluation of Corneal Higher-Order Aberrations Before and After LASIK
Brief Title: Scheimpflug Versus Placido-disc System in Evaluation of Corneal Higher-Order Aberrations
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naglaa Mostafa Abdelhafez Abdelmohsen, Assistant lecturer, Assiut University
Other Study IDs: Corneal HOA
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Corneal Higher-order Aberrations
Keywords: higher-order aberrations; Pentacam; Topolyzer; LASIK

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: placido-based topographer (wavelight allegro topolyzer vario) and scheimpflug -based (Oculus Pentacam ) — An informed written consent will be obtained from all patients that will be included in this study. Patients in this study will undergo pentacam and topolyzer examination to asses corneal high order aberrations before LASIK procedure.
  Patients will be assigned to undergo LASIK. Follow up pentacam and topolyzer examination will be done 3 months after LASIK.

SUMMARY:
Aim of work:

To assess the agreement between placido-based topographer (wavelight allegro topolyzer vario) and scheimpflug -based (Oculus Pentacam ) regard measuring corneal higher order aberrations before and after LASIK.

DETAILED DESCRIPTION:
Higher-order aberrations (HOAs) are small optical irregularities of the eye, which can have an impact on the quality of the retinal image. In contrast to lower order aberrations, these errors cannot be corrected with regular spectacles and most contact lenses. Additionally, HOAs are responsible for an array of visual symptoms including dysphotopsia, glare, as well as a reduction in contrast sensitivity. The cornea accounts for approximately 90% of ocular aberrations.Advances and breakthroughs in wavefront aberration measurement technology can help clinicians to better understand and manage corneal higher-order aberrations (HOAs), especially for the preoperative planning of corneal refractive surgery and cataract surgery.A recent study has shown that corneal HOAs can be a sensitive parameter to differentiate early keratoconus from normal eyes. Furthermore, corneal aberrations have been widely used to evaluate dry eye and orthokeratology.LASIK surgery is widely used in the correction of refractive errors It is well known that LASIK surgery induces high-order aberrations (HOA) .The main eye element involved in the generation of such aberrations is the first corneal surface. Currently, devices based on Placido-disc, Hartmann- Shack, ray tracing, or Scheimpflug are routinely used in clinical aberration measurement. Of which Pentacam is one of common instruments that can only measure corneal aberration (including anterior and posterior corneal surface) based on Scheimpflug technology. Also Allegro Topolyzer is a Placido-based topographer that can measure anterior corneal higher order aberrations (HOAs). A better understanding of the agreement of device measurements can provide clinicians with useful information for measuring, correcting, and monitoring aberrations around refractive and cataract surgery. Investigators , therefore, aimed to study the agreement between the two instruments in anterior corneal aberration measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractive errors from +6 diopters to -8 diopters sphere and up to -6diopters cylinder.

Exclusion Criteria:

* Patients with systemic diseases such as diabetes.
* keratoconus or keratoconus suspect, amblyopic eyes.
* Patients with best corrected visual acuity (BCVA) not achieving 20/25.
* glucoma
* Previous ocular surgeries or trauma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who will undergo LASIK
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Agreement between placido-based topographer (wavelight allegro topolyzer vario) and scheimpflug -based (pentacam) | Before LASIK and 3 months after LASIK
  Agreement between placido-based topographer (wavelight allegro topolyzer vario) and scheimpflug -based (pentacam) regard measuring corneal high order aberrations before and after LASIK.

SECONDARY OUTCOMES:
Changes in high order aberrations after LASIK. | Before LASIK and 3 months after LASIK
  Changes in high order aberrations after LASIK using pentacam and topolyzer

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A Ali, Professor, Study Director — Assiut University; Khaled A Mohamed, Assistant prof, Study Director — Assiut University; Islam M Goda, Lecturer, Study Director — Assiut University
Locations (1):
- Naglaa Moustafa, Asyut, Egypt

REFERENCES:
- [Background] Salman A, Kailani O, Ghabra M, Omran R, Darwish TR, Shaaban R, Ibrahim H, Alhaji H, Khalil H. Corneal higher order aberrations by Sirius topography and their relation to different refractive errors. BMC Ophthalmol. 2023 Mar 16;23(1):104. doi: 10.1186/s12886-023-02841-4. PMID 36927406
- [Background] Little JA, McCullough SJ, Breslin KM, Saunders KJ. Higher order ocular aberrations and their relation to refractive error and ocular biometry in children. Invest Ophthalmol Vis Sci. 2014 Jul 15;55(8):4791-800. doi: 10.1167/iovs.13-13533. PMID 25028356
- [Background] Ning R, Huang X, Jin Y, Lei CS, Ma X, Xu S, Xiahou J, Savini G, Schiano-Lomoriello D, Wang X, Zhou X, Huang J. Corneal Higher-Order Aberrations Measurements: Precision of SD-OCT/Placido Topography and Comparison with a Scheimpflug/Placido Topography in Eyes After Small-Incision Lenticule Extraction. Ophthalmol Ther. 2023 Jun;12(3):1595-1610. doi: 10.1007/s40123-023-00693-1. Epub 2023 Mar 2. PMID 36862309
- [Background] Lou W, Du W, Jin H, Hu Y. Comparison of anterior corneal aberrations measured by Scheimpflug and Placido Disc System for myopes. BMC Ophthalmol. 2022 Dec 28;22(1):512. doi: 10.1186/s12886-022-02753-9. PMID 36578031
- [Background] Miret JJ, Rojas E, Camps VJ, Garcia C, Caballero MT, Martín B, et al. Understanding the Real Effect of the High-Order Aberrations after Myopic Femto-Lasik. Optics. 2022;3(4):384-99.
- [Background] Mai EL, Chang CK, Lee CY, Lian IB, Chao CC. Higher-Order Aberrations of Topography-Guided LASIK and Wavefront-Optimized LASIK in High- and Low-Myopic Eyes: A Non-Randomized Controlled Trial. J Pers Med. 2023 Feb 24;13(3):399. doi: 10.3390/jpm13030399. PMID 36983581
- [Background] Piccinini AL, Golan O, Hafezi F, Randleman JB. Higher-order aberration measurements: Comparison between Scheimpflug and dual Scheimpflug-Placido technology in normal eyes. J Cataract Refract Surg. 2019 Apr;45(4):490-494. doi: 10.1016/j.jcrs.2018.11.015. Epub 2019 Jan 31. PMID 30713018
- [Background] Ortiz-Toquero S, Rodriguez G, de Juan V, Martin R. Repeatability of Wavefront Aberration Measurements With a Placido-Based Topographer in Normal and Keratoconic Eyes. J Refract Surg. 2016 May 1;32(5):338-44. doi: 10.3928/1081597X-20160121-04. PMID 27163620